CLINICAL TRIAL: NCT01717625
Title: The Efficacy and Safety of Montelukast Sodium in the Prevention of Bronchopulmonary Dysplasia
Acronym: BPD
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Ajou University School of Medicine (Other)
Collaborators: Severance Hospital (Other); Seoul National University Hospital (Other); Gangnam Severance Hospital (Other); Korea University (Other)
Responsible Party: Principal Investigator, Lee Janghoon, Assistant professor, Ajou University School of Medicine
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: AJIRB-MED-CT2-11-242
Record Dates: First submitted 2012-10-26; First posted 2012-10-30 (Estimated); Last update posted 2015-02-10 (Estimated); Status verified 2015-02

CONDITIONS: Premature Birth; Infant, Very Low Birth Weight; Bronchopulmonary Dysplasia
Keywords: montelukast; BPD; singulair; prematurity
MeSH Terms: conditions — Premature Birth; Bronchopulmonary Dysplasia | interventions — montelukast

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Montelukast (Experimental): montelukast sodium
  * dosage
    * < 1000g : 0.5 mg/D QD
    * 1000g~1500g : 1.0 mg/D QD
    * 1500g~2000g : 1.5 mg/D QD
    * > 2000g : 2mg/D QD
  * medication period : to discharge or GA 36wks
  Interventions: Drug: Montelukast
- Control (No Intervention): Standard treatment of BPD and preterm infants

INTERVENTIONS:
Drug: Montelukast — a leukotriene D4 receptor antagonist; sodium salt is the active compound; structure in first source
  Other Names: Singulair
  Arms: Montelukast

SUMMARY:
This study is multicentered, prospective, randomized, opened, parallel, intervention study.

The aim of this study is to evaluate the efficacy and safety of Montelukast sodium in the prevention of bronchopulmonary dysplasia (BPD) in preterm infant, below 32weeks gestational age.

The investigators evaluate the first effectiveness through the morbidity and mortality of bronchopulmonary dysplasia. And then, the investigators evaluate the second effectiveness through the oxygen index, the usage of mechanical ventilator about taking medicine after 2 Weeks, Oxygen Utilization After 4 Weeks, Proinflammatory Cytokine through the bronchial lavage fluid.

ELIGIBILITY:
Inclusion Criteria:

* Preterm infants born at less than 32 weeks
* Birth 14 days after, oxygen or artificial ventilation who are using patient
* more than 20cal/kg/d by enteral feeding
* written consent of the parents

Exclusion Criteria:

* congenital anomaly
* cardiovascular collapse
* investigator's opinion

Ages: 2 Weeks to 10 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 72 (Actual)
Dates: Start 2011-11; Primary Completion 2013-10 (Actual); Study Completion 2013-10 (Actual)

PRIMARY OUTCOMES:
Incidence of moderate to severe BPD or mortality | corrected gestational age
  At corrected gestational age 36 weeks, to compare the incidence of moderate to severe BPD or mortality

SECONDARY OUTCOMES:
Oxygen Index. Use of mechanical ventilation, oxygen, systemic steroid. Weight gain, adverse event | 1, 2, 4 weeks since starting study

CONTACTS AND LOCATIONS:
Overall Officials: Moonsung Park, professor, Study Chair — Ajou University Medical Center
Locations (1):
- Ajou university medical center, Suwon, Woncheon-dong, Yeongtong-gu,, South Korea